CLINICAL TRIAL: NCT02792348
Title: Change of Urinary Metabolic Profile Secondary to a Congenital Urine Flow Impairment (UFI) by Nuclear Magnetic Resonance (NMR) and Metabolomics Analysis
Acronym: ACEU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50720
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Congenital Urine Flow Impairment
Keywords: congenital urine flow impairment; urinary metabolomics profile; Nuclear Magnetic Resonance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — De-identified and study coded urine samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- children with congenital urine flow impairment: this group contain children with an unilateral urinary tract dilatation diagnosed by prenatal ultrasonography
  Interventions: Other: Laboratory biomarker analysis on urine sample
- control group: this group contains children, between 1 and 3 months of age, without nephrological or urological anomaly
  Interventions: Other: Laboratory biomarker analysis on urine sample

INTERVENTIONS:
Other: Laboratory biomarker analysis on urine sample — Archived urine samples are analyzed for specific metabolite patterns by nuclear magnetic resonance

SUMMARY:
For the new-born, diagnosis and prognosis of congenital urine flow impairment (UFI) are difficult to confirm only with morphological examination (ultrasonography, intravenous pyelography) and functional examination (dynamic renal scan MAG3). Only the test of time allows the post confirmation of a significant UFI requiring a surgery. This meant that the actual therapeutic indications are imperfect by the absence of an "absolute" endpoint for UFI.

The objective of the study is to characterize the urinary metabolomics profile of new born with renal pelvis and/or ureters tract dilatation (suspicion of pelvi-ureteric junction anomalies, primary megaureter and vesico-ureteric reflux), detected by prenatal ultrasonography, by Nuclear Magnetic Resonance (NMR) and metabolomics analysis. This characterization will allow the identification of statistically significant metabolomics markers for the diagnosis and prognosis of a favourable evolution of the anomaly. The evolution with time of these metabolomics profiles will also considered.

ELIGIBILITY:
* Inclusion Criteria - UFI group:

  * Newborns or infants between 1 and 3 months of age,
  * who present an upper urinary tract dilatation detected on prenatal ultrasound scanning, and confirmed with a postnatal sonographic investigation between D4 and D10 of life showing a renal pelvis with an anteroposterior diameter > 10 mm and/or an ureters > 6 mm,
  * Written, informed consent obtained from the 2 parents
* Inclusion Criteria - control group:

  * Newborns or infants between 1 and 3 months of age,
  * Written, informed consent obtained from the 2 parents
* Non-inclusion Criteria - UFI group:

  * urological associated anomaly: bladder dysfunction, solitary kidney, bilateral pathology,
  * Absence of parents consent
* Non-inclusion Criteria - control group:

  * Nephrologic or urological anomaly
  * Previous medical conditions or prior surgery; except minor surgery (inguinal hernia, umbilical hernia, hypertrophic pyloric stenosis…..)
  * Absence of parents consent

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All patients (newborns or infants between 1 and 3 months of age) will be enrolled outpatient uro-visceral service of HFME hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-02; Primary Completion 2015-01 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
NMR identification of urinary metabolomics markers for diagnosis and prognosis of UFI (suspicion of pelvi-ureteric junction anomalies, primary megaureter and vesico-ureteric reflux) detected in prenatal ultrasonography. | Urine samples of patients will be collected at recruitment time (Day 0).
  Urine will be stored at _80 _C before acquisition of the NMR data. Urine samples will be thawed at room temperature before use. 400µL of supernatant will be diluted with 200 µL of a buffer solution Na2HPO4/NaH2PO4 (pH = 7.4; 20% D2O/H2O v.v, internal reference: 3-(trimethylsilyl)propionic,2-2-3-3-d4 acid) in Eppendorf tubes. Each sample will be centrifuged for 5 min at 4°C at 12,000 g. Finally, 550 µL will be transferred into 5 mm NMR tubes for analysis. Standard 1H 1D NMR pulse sequences, NOESY and CPMG with water presaturation, will be applied on each sample to obtain corresponding metabolic profiles. In addition, 2D NMR experiments (1H-1H TOCSY or 1H-13C HSQC, and 1H J-Resolved) will be recorded to achieve structural assignment of the metabolic signals.

SECONDARY OUTCOMES:
change of the urinary metabolomics profile change of UFI (pelvi-ureteric junction anomalies, primary megaureter and vesico-ureteric reflux) during the follow-up. | Urine samples of patients will be collected at the follow-up visits between 9 and 12 months of age (M9-M12).
  Urine will be stored at _80 _C before acquisition of the NMR data. Urine samples will be thawed at room temperature before use. 400µL of supernatant will be diluted with 200 µL of a buffer solution Na2HPO4/NaH2PO4 (pH = 7.4; 20% D2O/H2O v.v, internal reference: 3-(trimethylsilyl)propionic,2-2-3-3-d4 acid) in Eppendorf tubes. Each sample will be centrifuged for 5 min at 4°C at 12,000 g. Finally, 550 µL will be transferred into 5 mm NMR tubes for analysis. Standard 1H 1D NMR pulse sequences, NOESY and CPMG with water presaturation, will be applied on each sample to obtain corresponding metabolic profiles. In addition, 2D NMR experiments (1H-1H TOCSY or 1H-13C HSQC, and 1H J-Resolved) will be recorded to achieve structural assignment of the metabolic signals.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de LYon - Hôpital Femme Mère Enfant, Bron, France